CLINICAL TRIAL: NCT06640660
Title: Investigating Visuo-spatial Abilities and Psychological Effects in West Nile and Multiple Sclerosis Patients with a Focus on a Possible Rehabilitation Protocol
Acronym: Visuomind
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Camillo, Venezia, Italy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022.11
Record Dates: First submitted 2024-03-07; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Multiple Sclerosis; West Nile Virus
Keywords: neurological patients; cognitive training; neuropsychology
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MindLenses Group (Experimental): The group will undergo 10 sessions (2 weeks) of a treatment combining prismatic adaptation (PA) and serious games (SG) for cognitive training, using the Mindlenses Professional device. In each session, the PA procedure will be performed, followed by approximately 30 minutes of SG. SG will be focused on attention, executive functions and language.
  Interventions: Device: Mindlenses Professional
- Control Group (Active Comparator): The group will perform 2 weeks of the standard cognitive training offered by IRCCS San Camillo Hospital.
  Interventions: Behavioral: Conventional rehabilitation

INTERVENTIONS:
Device: Mindlenses Professional — MindLenses professional's device combines the prismatic adaptation (PA) procedure with the administration of serious games (SG) for cognitive training using a tablet
  Arms: MindLenses Group
Behavioral: Conventional rehabilitation — Conventional rehabilition consists in computerized exercises focused on the main cognitive domains
  Arms: Control Group

SUMMARY:
The study aims to investigate visuospatial abilities and psychological outcomes in patients with multiple scleroris (MS) and patients with West Nile virus infection (vWN). Patients will undergo a specific neuropsychological and psychological evaluation. Afterwards, patients will receive 10 sessions of cognitive training integrating digital exercises and prismatic lenses. At the end of the treatment, patients will be re-evaluated to explore for potential changes in the cognitive and psychological profile.

DETAILED DESCRIPTION:
Over time, the literature has investigated the impairment of cognitive and psychological aspects in patients with vWN and MS, due to the fact that both conditions can affect normal cognitive functioning.

As far as VWN is concerned, most cases in humans are asymptomatic, while about 20% of infected subjects develop a disease defined as West Nile fever, characterized by symptoms such as fever, headache, muscle pain, possible skin rashes, and lymphadenopathy. Less than 1% of infected people develop a form of the virus defined as neuro-invasive, which can manifest itself through encephalitis, meningitis, and flaccid paralysis. From a cognitive point of view, following the development of the disease, the difficulties mainly reported by patients concern memory loss, the decrease in motor skills, the onset of depression, and the inability to carry out the activities of daily life as before the illness. Furthermore, deficits in attention and executive functions have been identified through the use of neuropsychological tests. The few studies present in the literature that have investigated the state of the cognitive system in patients with vWN often do not agree with the definition of a characteristic pattern. Therefore, a short pilot was carried out to evaluate cognitive deficits in patients with VWN outcomes currently hospitalized at the San Camillo IRCCS. From this pilot, it emerged that the main difficulties concern the attentional, executive, and visuospatial functions.

Even in MS, a chronic inflammatory, demyelinating, and degenerative disease of the central nervous system, cognitive deficits are often present, especially in patients with the Relapsing Remitting or Progressive form. Furthermore, more than 50% of patients experience depression. Cognitive impairment can affect specific functions or be severe and widespread, depending on the location of the brain lesions caused by the disease. In any case, the most affected cognitive functions are attention and information processing speed, short and long-term memory in its explicit subcomponent and prospective memory, executive functions, language, and visuospatial functions. However, as far as the latter are concerned, on the one hand, there are few studies that have investigated the visuospatial component in MS; on the other, these studies report inconsistent results, also due to the heterogeneity in the applied tests and in the terminology used to define these deficits. In these studies, in fact, the difference between visuospatial and visuo-perceptive deficits is not always clear, with a consequent, sometimes non-specific use of the relative tests.

Since the literature has not investigated the visuo-spatial deficit in vWN disease, further studies are needed to explore this disorder in patients with vWN infection outcomes and with MS for the role that this function plays in daily life. In fact, visuo-spatial skills allow the person to relate correctly with the surrounding environment, orienting himself and regulating his own behavior according to it. A deficit at this level compromises both personal and professional quality of life.

The present study arises from the need to investigate more fully the visuo-spatial component in patients with vWN infection outcomes and with MS and aims to evaluate the effectiveness of an innovative tool for its treatment.

The procedure to be used involves the use of prismatic lenses since their efficacy in the rehabilitation of visuo-spatial deficits has been demonstrated.

To this end, the treatment administered will be Mindlenses Professional, a cognitive rehabilitation tool that allows to combine the traditional prismatic adaptation procedure with serious games delivered through a tablet and aimed at rehabilitating other cognitive functions such as attention and executive functions. Several researchers have begun to use prismatic lenses as a non-invasive neuromodulation tool: the prismatic adaptation process would, in fact, allow to act on cortical excitability, in particular by increasing the excitability of the frontal and parietal cortices ipsilaterally to the lens-induced deviation.

Mindlenses Professional could, therefore, prove to be an effective tool for the rehabilitation of patients with outcomes of vWN infection and MS who also have deficits in visuospatial functions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of: Multiple Scleroris OR vWN infection ascertained by laboratory analysis and received no later than twelve months prior to the date of hospitalization
* preserved use of at least one hand
* normal or corrected to normal vision

Exclusion Criteria:

* history of psychiatric and/or concurrent neurological diseases
* inability to provide informed consent,
* impaired comprehension of oral instructions,

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-09-21 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Measure of changes in cognitive performance after the treatment | At baseline and after 2 weeks (post-intervention)
  Cognitive performances will be assessed by a full neuropsychological battery encompassing the main cognitive domain, such as memory, attention, executive function, language, visuospatial abilities. Specific neuropsychological tests will be defined on the basis of the specific neurological population.
  Raw scores at each test and scale will be converted in z-scores based on each test/scale normative data. Z-scores will be averaged to calculate composite scores specific for each cognitive domain and for motor functioning. In detail, the composite scores will be the following: general cognitive functioning, attention, executive function, short-term memory, long-term memory, visuospatial abilities, language.

SECONDARY OUTCOMES:
Measure of changes in psychological aspects after the treatment | At baseline and after 2 weeks (post-intervention)
  Psychological measures will be administered to investigate the presence of anxiety and depression in each patient.
  Questionnaires will be scored based on published norms.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Camillo Hospital, Lido, Venezia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bracco M, Mangano GR, Turriziani P, Smirni D, Oliveri M. Combining tDCS with prismatic adaptation for non-invasive neuromodulation of the motor cortex. Neuropsychologia. 2017 Jul 1;101:30-38. doi: 10.1016/j.neuropsychologia.2017.05.006. Epub 2017 May 6. PMID 28487249
- [Background] Carson PJ, Konewko P, Wold KS, Mariani P, Goli S, Bergloff P, Crosby RD. Long-term clinical and neuropsychological outcomes of West Nile virus infection. Clin Infect Dis. 2006 Sep 15;43(6):723-30. doi: 10.1086/506939. Epub 2006 Aug 10. PMID 16912946
- [Background] Chiaravalloti ND, DeLuca J, Moore NB, Ricker JH. Treating learning impairments improves memory performance in multiple sclerosis: a randomized clinical trial. Mult Scler. 2005 Feb;11(1):58-68. doi: 10.1191/1352458505ms1118oa. PMID 15732268
- [Background] Chiaravalloti ND, DeLuca J. Cognitive impairment in multiple sclerosis. Lancet Neurol. 2008 Dec;7(12):1139-51. doi: 10.1016/S1474-4422(08)70259-X. PMID 19007738
- [Background] Hayes EB, Sejvar JJ, Zaki SR, Lanciotti RS, Bode AV, Campbell GL. Virology, pathology, and clinical manifestations of West Nile virus disease. Emerg Infect Dis. 2005 Aug;11(8):1174-9. doi: 10.3201/eid1108.050289b. PMID 16102303
- [Background] Magnani B, Caltagirone C, Oliveri M. Prismatic adaptation as a novel tool to directionally modulate motor cortex excitability: evidence from paired-pulse TMS. Brain Stimul. 2014 Jul-Aug;7(4):573-9. doi: 10.1016/j.brs.2014.03.005. Epub 2014 Apr 13. PMID 24934876
- [Background] Pisella L, Rode G, Farne A, Tilikete C, Rossetti Y. Prism adaptation in the rehabilitation of patients with visuo-spatial cognitive disorders. Curr Opin Neurol. 2006 Dec;19(6):534-42. doi: 10.1097/WCO.0b013e328010924b. PMID 17102690
- [Background] Rao SM, Leo GJ, Bernardin L, Unverzagt F. Cognitive dysfunction in multiple sclerosis. I. Frequency, patterns, and prediction. Neurology. 1991 May;41(5):685-91. doi: 10.1212/wnl.41.5.685. PMID 2027484